CLINICAL TRIAL: NCT02067377
Title: A Randomized, Double Blinded, Placebo-controlled Pilot Study of Serum Bovine Immunoglobulin (SBI) for Cachexia in Patients With Advanced COPD
Brief Title: Efficacy of Serum Bovine Immunoglobulin in Improving Nutritional Status in Advanced COPD
Acronym: SBI for COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Entera Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000027289
Record Dates: First submitted 2014-02-06; First posted 2014-02-20 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Advanced COPD (GOLD Stage 3 or 4) With Cachexia
Keywords: GOLD, COPD, cachexia, BMI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cachexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- inactive powder substance (Placebo Comparator): inactive powder substance by mouth twice a day for 6 months
  Interventions: Dietary Supplement: Placebo (for serum bovine immunoglobulin)
- serum bovine immunoglobulin (SBI) medical food (Experimental): SBI medical food 5 gr powder substance by mouth twice a day for 6 months
  Interventions: Dietary Supplement: Serum bovine immunoglobulin (SBI) medical food
- serum bovine immunoglobulin (SBI) medicalfood (Experimental): SBI medical food 10 gr powder substance by mouth twice a day for 6 months
  Interventions: Dietary Supplement: Serum bovine immunoglobulin (SBI) medical food

INTERVENTIONS:
Dietary Supplement: Serum bovine immunoglobulin (SBI) medical food — Serum bovine immunoglobulin (SBI) is an FDA regulated, orally administered prescription medical food intended for the nutritional management of patients who are unable to absorb necessary nutrients as a result of therapeutic or chronic medical problems.
  Arms: serum bovine immunoglobulin (SBI) medical food; serum bovine immunoglobulin (SBI) medicalfood
Dietary Supplement: Placebo (for serum bovine immunoglobulin)
  Arms: inactive powder substance

SUMMARY:
This study will evaluate the use of a medical food, oral serum-derived bovine immunoglobulin/protein isolate (SBI), in helping patients with advanced COPD with cachexia (a wasting syndrome) improve their nutritional status and gain weight. The medical food is in powder form and is mixed with a liquid such as water or orange juice and consumed by swallowing. The primary hypothesis is that SBI protein isolate (SBI) will improve the nutritional status of cachexic patients with advanced stages of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age between age 30 and 80 at Baseline Visit
* Diagnosed with 2012 spirometric COPD GOLD Stage 3 (FEV1/FVC ratio <0.70, FEV1 30-49% of normal) or GOLD Stage 4 (FEV1/FVC <0.70, FEV1 <30% of normal or FEV1<50% of normal with chronic respiratory failure present)
* Able to tolerate and willing to undergo study procedures
* Body Mass Index below 21
* Signed Informed Consent

Exclusion Criteria:

* History of comorbid condition severe enough to significantly impact 6 months outcomes
* Current substance abuse, including tobacco, alcohol and illicit drugs
* Diagnosis of unstable cardiovascular disease including myocardial infarction in the past 6 weeks, uncontrolled congestive heart failure, or uncontrolled arrhythmia
* Dementia or other cognitive dysfunction which in the opinion of the investigator would prevent the participant from consenting to the study or completing study procedures
* Active pulmonary infection with tuberculosis
* Non-COPD obstructive lung disease (various bronchiolitides, sarcoidosis, LAM, histiocytosis X) or parenchymal lung disease, pulmonary vascular disease, pleural disease, severe kyphoscoliosis, neuromuscular weakness, or other cardiovascular and pulmonary disease, that limit the interpretability of the pulmonary function measures
* Prior significant difficulties with pulmonary function testing
* Hypersensitivity to or intolerance of albuterol sulfate or ipratropium bromide or propellants or excipients of the inhalers, or to beef
* History of lung or other organ transplant
* Currently taking >20mg of prednisone or equivalent systemic corticosteroid
* Currently taking any immunosuppressive agent
* History of lung cancer or any cancer that spread to multiple locations in the body
* Known HIV/AIDS infection
* History of or current exposure to chemotherapy or radiation treatments that, in the opinion of the investigator, limits the interpretability of the pulmonary function measures.
* Current or planned pregnancy within the study course.
* Currently institutionalized (e.g., prisons, long-term care facilities)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The subtracted differences in BMI, body fat measurement, and grip strength between participants receiving SBI or placebo at baseline and 6 months. | 6 months

SECONDARY OUTCOMES:
The subtracted differences between FEV1 and COPD Assessment Test scores in patients receiving SBI or placebo at baseline and 6 months. | 6 months

OTHER OUTCOMES:
The subtracted differences in swallowing-associated laryngeal Penetration Aspiration Scale (PAS) in patients receiving SBI or placebo at baseline and 6 months. | 6 months
The subtracted differences in mean serum TNF-alpha and IL-6 concentrations between participants receiving SBI or placebo at baseline and 6 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Luca Paoletti, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States